CLINICAL TRIAL: NCT04755426
Title: Understanding Patient Goals and Preferences to Facilitate Shared Decision Making for Symptomatic Aortic Stenosis
Status: Completed | Type: Observational
Sponsor: Shared Decision Making Resources (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Nananda Col, Founder, Shared Decision Making Resources
Other Study IDs: HCP-8243002
Record Dates: First submitted 2021-02-06; First posted 2021-02-16 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Aortic Stenosis Symptomatic
Keywords: Shared decision making; Preference assessment; Values clarification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with severe aortic stenosis: Adults with severe aortic stenosis who either have faced or are facing a decision about valve replacement (depending on the phase of the research)
  Interventions: Behavioral: AVITA--Aortic Valve Improved Treatment Approaches
- Health care providers: HCPs who guide decisions about managing AS, including interventional cardiologists, cardiac surgeons and advanced practice providers (APPs), including nurse practitioners and physician assistants.
  Interventions: Behavioral: AVITA--Aortic Valve Improved Treatment Approaches

INTERVENTIONS:
Behavioral: AVITA--Aortic Valve Improved Treatment Approaches — AVITA is an interactive shared decision making tool that helps patients clarify their treatment goals and preferences and communicate those preferences to their valve specialist.
  Other Names: Values Clarification Tool; Online learning tool; Shared decision making tool

SUMMARY:
The overall goal of this study is to develop and validate a preference assessment tool for patients who have severe aortic stenosis and are contemplating their treatment options. The first part of the study focuses on understanding the treatment goals and treatment features that matter most to patients who have already made the decision. The investigators use mixed methods (nominal group technique, card sorting) to elicit, prioritize, and organize these patient preferences into a "cognitive map". Based on those findings, the investigators design a preference tool and then pre-test the tool with patients and healthcare providers.

DETAILED DESCRIPTION:
The investigators are conducting a 4-phase phase mixed methods study involving nominal group technique (NGT), with patients driving the identification and categorization of preferences regarding treatment options for symptomatic AS. Participants include adults with a history of symptomatic AS and HCPs who guide decisions about managing AS, including interventional cardiologists, cardiac surgeons and advanced practice providers (APPs), including nurse practitioners and physician assistants.

The initial phases of the study (generating patient goals and preferences through NGTs) targets diverse patients with a history of severe Aortic Stenosis (AS) who have previously made the decision regarding treatment choices. This will include patients who have undergone Surgical aortic valve replacement (SAVR), Transcatheter aortic valve replacement (TAVR), or who elected palliative care with or without balloon valvuloplasty. The subsequent phases will include patients with AS who are currently facing a decision with regard to treatment.

Phase 1: Identify and prioritize patient a) goals and b) preferences for treatment. The nominal group technique (NGT) will be used to identify and prioritize patient-centered outcomes related to treatment goals and treatment features. Both in-person and online NGT groups, with 5-9 patients each, will be conducted to maximize the representativeness of the sample (6-8 NGTs). Planning for 4 NGT's per question (8 total), including a minimum of 2 in-person NGTs (and the remaining conducted either in-person or online, depending on which approach better enables recruitment needs. Each NGT has between 5 and 9 patients. A separate parallel process will be done for each NGT question including a) goals and b) preferences for treatment attributes to limit patient burden for each portion of the study.

Phase 2: Categorize patient a) goals and b) preferences for treatment through cognitive mapping. Following identification and prioritization of patient-generated goals and preferences, 25-50 patients across the three sites will participate online in "card sorting" activities that will be used to organize these prioritized lists into clusters (domains), using Multidimensional Scaling (MDS) and Hierarchical Cluster Analysis (HCA) to analyze the data. A parallel process will be done for each cognitive map including a) goals and b) preferences for treatment.

Phase 3: Based on patient-defined goals and preferences for the treatment of AS, develop the preference assessment tool. The patient-identified goals and preferences will serve as the core of the preference tool. The investigators will draw from a validated SDM template to summarize and communicate patient preferences to their HCPs. An early prototype will be developed, and subsequent usability testing with patients with a history of severe AS will refine the tool. The prototype that will be used is available at: https://tinyurl.com/WhatMattersMS

Phase 4: Pilot test the preference assessment tool using 20-25 patient-HCP pairs to compare HCPs' prediction of patient preferences to actual patient preferences, among those patients who have not yet received treatment for their AS. Before each clinical encounter, each HCP will be asked to infer their patient's top 1-3 treatment goals and preferences. Patients will have interacted with the preference assessment tool independently before the clinical appointment, which will have assessed and summarized their goals and preferences. After the HCP has entered his/her inferred patient treatment goals, he/she will be shown the patient's actual treatment goals and preferences. Analyses will compare the correspondence between the patient and HCP preferences (using Kappa statistic). Additionally, the outcomes below will be assessed in preparation for the subsequent national validation study.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic aortic stenosis (also known as severe aortic stenosis)
* English-speaking
* a patient of a participating HCP (for Phases 3 and 4)

Exclusion Criteria:

* 18 years of age or younger
* unable or unwilling to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient participants are identified through HCP advisers and patient advisers with access to a AS patient networks (Heart Valve Voice US), Women in Cardiology (private Facebook Group) using a purposive sampling design.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Shared Decision Making Process Scale | Within a day or 2 of meeting with their valve specialist to discuss treatment options
  A patient-reported measure of shared decision making with their clinician.

SECONDARY OUTCOMES:
Patient-identified preferences for treatment. | At baseline, while using the tool, and within a day or 2 of meeting with their valve specialist to discuss treatment options
  The treatment for aortic stenosis that the patient prefers (SAVR, TAVR, Medical Therapy, or undecided.
Healthcare providers' perceptions of their patient's preferences. | WIthin a few days of having an appointment with the patient who has interacted with the tool.
  The features (attributes) of their treatment options for aortic stenosis that matter most to the patient
CollaboRATE | Within a day or 2 of meeting with their valve specialist to discuss treatment options
  A short patient-reported measure of patient-provider communication
Knowledge (Subjective and objective) | At baseline, just after completing the tool, and within a day or 2 of meeting with their valve specialist.
  Multiple choice questions that assess perceived and actual knowledge about aortic stenosis and treatment options.

CONTACTS AND LOCATIONS:
Overall Officials: Nananda F Col, MD, MPH, Principal Investigator — Shared Decision Making Resources; Christina Fitzpatrick, MA, Study Director — Shared Decision Making Resources
Locations (1):
- Shared Decision Making Resources, Georgetown, Maine, United States

IPD SHARING:
Plan to Share IPD: Yes
All deidentified IPD. We plan to publish this information in scientific manuscripts.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the time of publication of our findings and for the following 2 years.
Access Criteria: Contact the study investigators.

REFERENCES:
- [Background] Col NF, Solomon AJ, Springmann V, Garbin CP, Ionete C, Pbert L, Alvarez E, Tierman B, Hopson A, Kutz C, Berrios Morales I, Griffin C, Phillips G, Ngo LH. Whose Preferences Matter? A Patient-Centered Approach for Eliciting Treatment Goals. Med Decis Making. 2018 Jan;38(1):44-55. doi: 10.1177/0272989X17724434. Epub 2017 Aug 14. PMID 28806143
- [Background] Col NF, Solomon AJ, Springmann V, Ionete C, Alvarez E, Tierman B, Kutz C, Morales IB, Griffin C, Ngo LH, Jones DE, Phillips G, Hopson A, Pbert L. Evaluation of a Novel Preference Assessment Tool for Patients with Multiple Sclerosis. Int J MS Care. 2018 Nov-Dec;20(6):260-267. doi: 10.7224/1537-2073.2017-021. PMID 30568563
- [Background] Witteman HO, Gavaruzzi T, Scherer LD, Pieterse AH, Fuhrel-Forbis A, Chipenda Dansokho S, Exe N, Kahn VC, Feldman-Stewart D, Col NF, Turgeon AF, Fagerlin A. Effects of Design Features of Explicit Values Clarification Methods: A Systematic Review. Med Decis Making. 2016 Aug;36(6):760-76. doi: 10.1177/0272989X16634085. Epub 2016 Apr 4. PMID 27044883
- [Background] Gallagher M, Hares T, Spencer J, Bradshaw C, Webb I. The nominal group technique: a research tool for general practice? Fam Pract. 1993 Mar;10(1):76-81. doi: 10.1093/fampra/10.1.76. PMID 8477899
- [Background] Stacey D, Legare F, Col NF, Bennett CL, Barry MJ, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L, Wu JH. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2014 Jan 28;(1):CD001431. doi: 10.1002/14651858.CD001431.pub4. PMID 24470076
- [Background] Col N, Hull S, Springmann V, Ngo L, Merritt E, Gold S, Sprintz M, Genova N, Nesin N, Tierman B, Sanfilippo F, Entel R, Pbert L. Improving patient-provider communication about chronic pain: development and feasibility testing of a shared decision-making tool. BMC Med Inform Decis Mak. 2020 Oct 17;20(1):267. doi: 10.1186/s12911-020-01279-8. PMID 33069228
- [Background] Col N, Alvarez E, Springmann V, Ionete C, Berrios Morales I, Solomon A, Kutz C, Griffin C, Tierman B, Livingston T, Patel M, van Leeuwen D, Ngo L, Pbert L. A Novel Tool to Improve Shared Decision Making and Adherence in Multiple Sclerosis: Development and Preliminary Testing. MDM Policy Pract. 2019 Oct 16;4(2):2381468319879134. doi: 10.1177/2381468319879134. eCollection 2019 Jul-Dec. PMID 31667351
- [Background] Lytvyn L, Guyatt GH, Manja V, Siemieniuk RA, Zhang Y, Agoritsas T, Vandvik PO. Patient values and preferences on transcatheter or surgical aortic valve replacement therapy for aortic stenosis: a systematic review. BMJ Open. 2016 Sep 29;6(9):e014327. doi: 10.1136/bmjopen-2016-014327. PMID 27687903
- [Background] Ho M, Saha A, McCleary KK, Levitan B, Christopher S, Zandlo K, Braithwaite RS, Hauber AB; Medical Device Innovation Consortium's Patient Centered Benefit-Risk Steering Committee. A Framework for Incorporating Patient Preferences Regarding Benefits and Risks into Regulatory Assessment of Medical Technologies. Value Health. 2016 Sep-Oct;19(6):746-750. doi: 10.1016/j.jval.2016.02.019. PMID 27712701
- [Background] Valentine KD, Vo H, Fowler FJ Jr, Brodney S, Barry MJ, Sepucha KR. Development and Evaluation of the Shared Decision Making Process Scale: A Short Patient-Reported Measure. Med Decis Making. 2021 Feb;41(2):108-119. doi: 10.1177/0272989X20977878. Epub 2020 Dec 15. PMID 33319648
- [Derived] Coylewright M, Otero D, Lindman BR, Levack MM, Horne A Jr, Ngo LH, Beaudry M, Col HV, Col NF. An interactive, online decision aid assessing patient goals and preferences for treatment of aortic stenosis to support physician-led shared decision-making: Early feasibility pilot study. PLoS One. 2024 May 21;19(5):e0302378. doi: 10.1371/journal.pone.0302378. eCollection 2024. PMID 38771808
- [Derived] Col NF, Otero D, Lindman BR, Horne A, Levack MM, Ngo L, Goodloe K, Strong S, Kaplan E, Beaudry M, Coylewright M. What matters most to patients with severe aortic stenosis when choosing treatment? Framing the conversation for shared decision making. PLoS One. 2022 Aug 11;17(8):e0270209. doi: 10.1371/journal.pone.0270209. eCollection 2022. PMID 35951553